CLINICAL TRIAL: NCT02945566
Title: STAR-TREC: Can We Save the Rectum by Watchful Waiting or TransAnal Surgery Following (chemo)Radiotherapy Versus Total Mesorectal Excision for Early REctal Cancer?
Brief Title: Can We Save the Rectum by Watchful Waiting or TransAnal Surgery Following (chemo)Radiotherapy Versus Total Mesorectal Excision for Early REctal Cancer?
Acronym: STAR-TREC
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_15-011; 2016-000862-49 (EudraCT Number)
Record Dates: First submitted 2016-07-25; First posted 2016-10-26 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Adenocarcinoma of the Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard TME surgery (Active Comparator): Radical total mesorectal excision
  Interventions: Procedure: Standard TME surgery
- Long course concurrent chemoradiation (Experimental): Capecitabine: 825 mg/m² orally, b.i.d., on radiotherapy days Radiotherapy: A dose of 50 Gy, applied to the primary tumour and surrounding mesorectum, in 25 fractions of 2 Gy, 5 days a week.
  Interventions: Drug: Long course concurrent chemoradiation with capecitabine and radiotherapy
- Short course radiotherapy (Experimental): A dose of 25Gy, applied, to the primary tumour and surrounding mesorectum in 5 fractions of 5 Gy, 5 days a week.
  Interventions: Radiation: Short course radiotherapy

INTERVENTIONS:
Procedure: Standard TME surgery — Total mesorectal excision
  Arms: Standard TME surgery
Drug: Long course concurrent chemoradiation with capecitabine and radiotherapy — Capecitabine 825 mg/m² orally, b.i.d., on radiotherapy days. Radiotherapy: A dose of 50 Gy, applied to the primary tumour and surrounding mesorectum, in 25 fractions of 2 Gy, 5 days a week.
  Other Names: Xeloda is the brand name for capecitabine
  Arms: Long course concurrent chemoradiation
Radiation: Short course radiotherapy — A dose of 25Gy, applied, to the primary tumour and surrounding mesorectum in 5 fractions of 5 Gy, 5 days a week.
  Arms: Short course radiotherapy

SUMMARY:
Bowel cancer is the second most common tumour with 41 000 new cases diagnosed annually in the UK, 447 000 across Europe and 1.36 million worldwide; of which one third are located in the rectum. Standard primary radical Total Mesorectal Excision (TME) surgery is an oncologically effective treatment for early stage rectal cancer. However, resection of a low rectal tumour requires a permanent stoma in approximately 10% of cases while many more patients have a temporary stoma, some of which are not reversed. Radical surgery, which evolved to treat locally advanced, symptomatic tumours, may not be the optimal method of treatment for early screen-detected tumours and an organ preserving strategy may generate significantly less morbidity without substantially compromising oncological outcomes.

STAR-TREC is a rolling phase II/III study. Phase II aimed to assess the feasibility of a large, multi-centre randomised trial comparing radical surgery versus two contrasting organ saving treatments followed by selective transanal microsurgery. Phase III will evaluate two contrasting organ preservation strategies in terms of organ preservation rates, toxicity (clinician and patient-reported) and Health-Related Quality of Life (HRQoL).

DETAILED DESCRIPTION:
The Phase II component of STAR-TREC (now completed) was a randomised, three arm (1:1:1) study using the following arms:

1. Standard TME surgery (control)
2. Organ saving treatments using:

   1. Long course concurrent chemoradiation:

      * Capecitabine: 825 mg/m² orally, b.d., on radiotherapy days
      * Radiotherapy: A dose of 50 Gy applied to the primary tumour and surrounding mesorectum in 25 fractions of 2 Gy, 5 days a week.
   2. Short course radiotherapy:

      * A dose of 25 Gy applied to the primary tumour and surrounding mesorectum in 5 fractions of 5 Gy, 5 days a week.

The phase III component of STAR_TREC is now open and has a partially randomised patient preference design where patients choose between organ saving treatment or standard surgery.

Those who prefer organ preservation will undergo randomisation 1:1 between:

1. Long course concurrent chemoradiation (as described above)
2. Short course radiotherapy (as described above)

Those who prefer standard surgery or have no preference, will undergo standard TME surgery without neoadjuvant radiotherapy treatment.

For organ-preserving strategies in phase II and III, clinical response to radiotherapy determines the next treatment step. Radiotherapy response is evaluated using clinical exam, endoscopy and MRI. The first assessment at 11-13 weeks (from radiotherapy start) using composite clinical, endoscopic and MRI based assessment will identify a minority of non-responders who should convert to TME surgery. Patients demonstrating a satisfactory radiotherapy response at 11-13 weeks will be reassessed by endoscopy at 16-20 weeks. Re-evaluation at 16-20 weeks determines if the STAR-TREC criteria for complete response (CR) are met. Patients who achieve CR may progress directly to active surveillance. Those who do not fulfil the criteria for CR will progress to excision biopsy with transanal endoscopic microsurgery (TEM).

The phase II component of the study aimed to evaluate the feasibility of accelerating patient recruitment from 2 per month, as attained in the previous TREC study, to 6 per month internationally over a two-year period.

The STAR-TREC phase III study will evaluate whether a CRT or SCRT organ preservation strategy leads to higher organ preservation rates and should become first line treatment for early rectal cancer.

This objective can be divided into two main questions:

1. Determine the optimal radiation schedule to achieve the highest rate of organ preservation
2. Determine the optimal radiation schedule to achieve the best quality of life after organ preservation

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the rectum
* MRI-defined ≤T3b (with ≤5mm of mesorectal invasion) rectal tumour or endorectal ultrasound-defined ≤uT3b rectal cancer (optional: in centres where high quality endorectal ultrasound (ERUS) is available or patient unable to tolerate MRI)
* MDT determines that all of the following treatment options are reasonable and feasible:

  --TME surgery, (b) CRT (c) SCRT d) TEM.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* For patients choosing organ preservation only:

  * If female and of childbearing potential, must:

    * Have a negative pregnancy test within 7 days prior to study entry
    * Agree to use adequate, medically approved, contraceptive precautions from trial entry until 6 months after the end of study treatment
  * If non-sterilised male male with a partner of childbearing potential, must:
  * Agree to use adequate, medically approved, contraceptive precautions from trial entry until 6 months after the end of study treatment
* Patient able and willing to provide written informed consent for the study

Exclusion Criteria:

* Concomitant or previous malignancies within 3 years prior to trial entry, except those that in the opinion of the MDT are unlikely to relapse within 3 years or lead to death within 5 years
* Unequivocal evidence of metastatic disease (includes resectable metastases)

  -- Patients with equivocal radiological lesions (e.g. retroperitoneal, liver, lung) that are not classified as M1 are eligible if agreed by MDT
* MRI node positive (≥N1, defined by protocol guidelines)

  -- Patients with equivocal radiological findings that are either classified as NX or N0 are eligible
* MRI extramural vascular invasion (mriEMVI) positive (defined by protocol guidelines)
* MRI defined mucinous tumour
* Mesorectal fascia threatened (≤1 mm on MRI or ERUS)
* Maximum tumour diameter > 40mm (either measured from everted edges on sagittal MRI or on ERUS)
* Tumour position anterior, above the peritoneal reflection on MRI or EUS
* No residual luminal tumour following endoscopic resection
* Contraindications to radiotherapy including previous pelvic radiotherapy
* Uncontrolled cardiorespiratory comorbidity (includes patients with inadequately controlled angina or myocardial infarction or arrhythmia within 6 months prior to trial entry)
* Known complete dihydropyrimidine dehydrogenase (DPYD) deficiency
* Known Gilbert's disease (hyperbilirubinaemia)
* Taking coumarin-derivative anticoagulants (e.g. warfarin) that cannot be discontinued at least 7 days prior to starting treatment or substituted by low molecular weight heparin
* Taking phenytoin or sorivudine or its chemically related anologues, such as brivudine, within 4 weeks of trial entry (see Section 8.3.5 for further details)
* Taking metronidazole at study entry
* Pregnant or lactating women
* History of severe and unexpected reactions to fluoropyrimidine therapy
* Age <16 years (UK), <18 years (other countries)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Phase II (Feasibility study) Primary Outcome: Recruitment Rate | 24 Months
  Measured at 12 and 24 months. Target recruitment rates are ≥4 and ≥6 patients randomised per month at 12 and 24 months respectively for total accrual of 120 international cases. Each individual country will attempt to exceed the minimum recruitment required to sustain phase III (UK 75, the Netherlands 75, Denmark 30). If recruitment is on target in year two then consideration will be given to an early application for transition to phase III with a funding application and a formal protocol amendment.
Phase III Primary Outcome: Organ Preservation | 30 Months from start day of (chemo)radiotherapy treatment.
  The primary endpoint of the STAR-TREC phase III study is the proportion of patients with successful organ preservation at 30 months from the start day of (chemo)radiotherapy treatment. This endpoint will be assessed for patients who prefer organ preservation and is defined as an in-situ rectum (includes patients subject to transanal local resection), no defunctioning stoma and an absence of active loco-regional cancer failure. The expected incidence of this outcome is approximately 60%.

SECONDARY OUTCOMES:
Phase II (Feasibility study): Core Endpoint - Funding | 12 Months
  Incidence of procurement of funding by one STAR-TREC international partner
Phase II (Feasibility study): Core Endpoint - International Recruitment | 12 Months
  Incidence of opening of STAR-TREC by one international partner
Phase II (Feasibility study): Core Endpoint - Efficacy | 12 Months
  Efficacy of organ preserving treatment arm on completion of phase II study: Is the organ saving rate more than 50% of patients with early stage rectal cancer at 12 months (following randomisation) achieved in the experimental arms? [Name of Measurement: Rate of organ saving >50% at 12 months; Unit of Measurement: no record of radical surgery at 12 months]
Phase II: Safety- Accuracy of MRI in predicting STAR-TREC eligibility | 24 Months
  MRI
  - Accuracy of MRI in predicting STAR-TREC eligibility (We will report the accuracy of MRI based patient selection according to each national standard, compared to the reference standard of post-operative histological staging. STAR-TREC will help develop international consensus in MRI reporting of mesorectal lymph node involvement by rectal cancer)
Phase II: Safety - 30 day Mortality | 30 days
  - Mortality
Phase II: Safety - 6 month Mortality | 6 Months
  - Mortality
Phase II: Safety - Surgical Morbidity | 36 Months
  - Surgical morbidity
Phase II: Safety - Tumour Recurrence/ Regrowth within Bowel Wall | 36 Months
  - Rate of tumour recurrence or regrowth within the bowel wall (experimental arm)
Phase II: Safety - Tumour Recurrence within Mesorectum | 36 Months
  - Rate of tumour recurrence within the mesorectum (experimental arm)
Phase II: Safety - Distant Metastasis | 36 Months
  - Rate of distant metastases
Phase II: Safety - Pelvic Failure | 36 Months
  - Pelvic failure rate: expressed as a sum of the following (i) unresectable pelvic tumour, (ii) cases requiring beyond TME surgery or (iii) tumour recurrence or regrowth ≤1mm from the circumferential surgical margin after TME surgery.
Phase II: Safety - Bowel | 36 Months
  Bowel dysfunction measured by EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] & C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items], LARS score [The Low Anterior Resection Syndrome score], and ICIQ-MLUTS/ICIQ-FLUTS [International Consultation on Incontinence Questionnaire Male/Female Lower Urinary Tract Symptoms Module]. Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomisation will be compared to baseline scores.
Phase II: Safety - Bladder | 36 Months
  Bladder dysfunction measured by EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] & C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items], LARS score [The Low Anterior Resection Syndrome score], and ICIQ-MLUTS/ICIQ-FLUTS [International Consultation on Incontinence Questionnaire Male/Female Lower Urinary Tract Symptoms Module]. Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomisation will be compared to baseline scores.
Phase II: Safety - Sexual dysfunction | 36 Months
  Sexual dysfunction measured by EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] & C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items], LARS score [The Low Anterior Resection Syndrome score], and ICIQ-MLUTS/ICIQ-FLUTS [International Consultation on Incontinence Questionnaire Male/Female Lower Urinary Tract Symptoms Module]. Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomisation will be compared to baseline scores.
Phase II: Efficacy - Stoma | 24 Months
  Additional outcome measures pertinent to the phase III study examining the efficacy of organ saving versus standard surgery will also be collected:
  - Proportion of patients with/ without a stoma at 30 days and one year
Phase II: Efficacy - Tumour Down-staging | 4.5 Months
  - Histopathological assessment of tumour down-staging following radiotherapy according to depth of tumour invasion and the incidence of other high-risk features in comparison to non-irradiated (control) group
Phase II: Efficacy - Active Monitoring | 4.5 Months
  - Proportion of patients identified by clinical and MRI assessment as suitable for active monitoring
Phase II: Efficacy - Conversion Rate | 36 Months
  - Conversion rates from organ saving to radical surgery
Phase II: Efficacy - Disease Survival | 36 Months
  - Disease free survival
Phase II: Efficacy - Health-related Quality of Life score | 3 months
  Quality of life measured by EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] & C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items], LARS score [The Low Anterior Resection Syndrome score], and ICIQ-MLUTS/ICIQ-FLUTS [International Consultation on Incontinence Questionnaire Male/Female Lower Urinary Tract Symptoms Module]. Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomisation will be compared to baseline scores.
Phase II: Efficacy - Health-related Quality of Life score | 12 Months
  Quality of life measured by EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] & C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items], LARS score [The Low Anterior Resection Syndrome score], and ICIQ-MLUTS/ICIQ-FLUTS [International Consultation on Incontinence Questionnaire Male/Female Lower Urinary Tract Symptoms Module]. Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomisation will be compared to baseline scores.
Phase II: Efficacy - Health-related Quality of Life score | 24 Months
  Quality of life measured by EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] & C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items], LARS score [The Low Anterior Resection Syndrome score], and ICIQ-MLUTS/ICIQ-FLUTS [International Consultation on Incontinence Questionnaire Male/Female Lower Urinary Tract Symptoms Module]. Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomisation will be compared to baseline scores.
Phase II: Efficacy - Health-related Quality of Life score | 36 Months
  Quality of life measured by EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] & C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items], LARS score [The Low Anterior Resection Syndrome score], and ICIQ-MLUTS/ICIQ-FLUTS [International Consultation on Incontinence Questionnaire Male/Female Lower Urinary Tract Symptoms Module]. Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomisation will be compared to baseline scores.
Phase II: Efficacy - Overall Survival | 36 Months
  - Overall survival
Phase III: For the randomised comparison between organ-preserving strategies | 30 days from start day of (chemo)radiotherapy treatment.
  Clinician-reported acute treatment related toxicity up to 30 days following completion of (chemo)radiotherapy
Phase III: Complete Response *For the randomised comparison between organ-preserving strategies | 30 months
  Proportion of patients with Complete Response to (chemo)radiation therapy
Phase III: For the randomised comparison between organ-preserving strategies - Local Excision | 20 weeks
  Proportion of patients undergoing transanal local excision
Phase III: For the randomised comparison between organ-preserving strategies - Organ Loss | Defined as the length of time from the start date of trial treatment until TME surgery
  Time to event of organ loss assessed for patients who prefer organ preservation
Phase III: For the randomised comparison between organ-preserving strategies - Non-Regrowth | 36 months
  Non-regrowth pelvic tumour control to 36 months; defined as the length of time from the start date of trial treatment until death (any cause) or development of unequivocal pelvic recurrence but not including patients who developed local regrowth which was resected with clear margins using standard TME surgery
Phase III: For the randomised comparison between organ-preserving strategies - Metastasis Free Survival | 36 months
  Metastasis free survival to 36 months; defined as the length of time from the start date of trial treatment until death (any cause) or detection of distant metastasis
Phase III: For the randomised comparison between organ-preserving strategies - Non-regrowth Disease Free Survival | 36 months
  Non-regrowth -disease free survival to 36 months; defined as the length of time from the start of trial treatment until death (any cause), detection of local pelvic recurrence or distant metastasis but not including patients who developed local regrowth which was resected with clear margins using standard TME surgery
Phase III: For the randomised comparison between organ-preserving strategies - Overall Survival | 60 months
  Overall survival to 60 months defined as the length of time from the start date of trial treatment until death (any cause)
Phase III: For analyses incorporating the non-randomised standard surgery comparator - Toxicity | 30 days
  Clinician-reported acute treatment related toxicity up to 30 days following completion of (chemo)radiotherapy or date of initial surgery
Phase III: For analyses incorporating the non-randomised standard surgery comparator - Non-regrowth Pelvic Tumour Control | 36 months
  Non-regrowth pelvic tumour control to 36 months; defined as the length of time from the start date of (chemo)radiotherapy or date of initial surgery until death (any cause) or development of unequivocal pelvic recurrence but not including patients who preferred organ preservation and developed local regrowth which was resected with clear margins using standard TME surgery
Phase III: For analyses incorporating the non-randomised standard surgery comparator - Metastasis Free Survival | 36 months
  Metastasis-free survival to 36 months; defined as the length of time from the start date of trial treatment or date of initial surgery until death (any cause) or detection of distant metastasis
Phase III: For analyses incorporating the non-randomised standard surgery comparator - Disease-free Survival | 36 months
  Disease-free survival to 36 months; defined as the length of time from the start date of trial treatment or date of initial surgery until death (any cause), detection of local pelvic recurrence or distant metastasis but not including patients who developed local regrowth which was resected with clear margins using standard TME surgery
Phase III: For analyses incorporating the non-randomised standard surgery comparator - Overall Survival | 60 months
  Overall survival to 60 months defined as the length of time from the start date of trial treatment or date of initial surgery until death (any cause))
Phase III: For analyses incorporating the non-randomised standard surgery comparator - Decision Regret | 24 months
  Decision regret at 24 months measured using the validated Decision regret scale questionnaire. The Decision Regret Scale is a 5-item Likert-type measure written to assess regret or remorse following a medical decision that takes less than 5 minutes to complete. High scores suggest high regret over a health care decision. Scores may be transformed to a scale of 0 (no regret) to 100 (high regret).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bach, MD, Principal Investigator — University Hospitals Birmingham
Locations (5):
- University Hospital UZ Leuven, Leuven, Belgium
- Odense University Hospital, Odense, Denmark
- Radboud University medical center, Nijmegen, Netherlands
- Region Stockholm, Onkologkliniken Södersjukhuset AB, Stockholm, Sweden
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Motamedi MAK, Mak NT, Brown CJ, Raval MJ, Karimuddin AA, Giustini D, Phang PT. Local versus radical surgery for early rectal cancer with or without neoadjuvant or adjuvant therapy. Cochrane Database Syst Rev. 2023 Jun 13;6(6):CD002198. doi: 10.1002/14651858.CD002198.pub3. PMID 37310167
- [Derived] Appelt AL, Kerkhof EM, Nyvang L, Harderwijk EC, Abbott NL, Teo M, Peters FP, Kronborg CJS, Spindler KG, Sebag-Montefiore D, Marijnen CAM; STAR-TREC collaborative group. Robust dose planning objectives for mesorectal radiotherapy of early stage rectal cancer - A multicentre dose planning study. Tech Innov Patient Support Radiat Oncol. 2019 Oct 15;11:14-21. doi: 10.1016/j.tipsro.2019.09.001. eCollection 2019 Sep. PMID 32095545
- [Derived] van den Ende RPJ, Peters FP, Harderwijk E, Rutten H, Bouwmans L, Berbee M, Canters RAM, Stoian G, Compagner K, Rozema T, de Smet M, Intven MPW, Tijssen RHN, Theuws J, van Haaren P, van Triest B, Eekhout D, Marijnen CAM, van der Heide UA, Kerkhof EM. Radiotherapy quality assurance for mesorectum treatment planning within the multi-center phase II STAR-TReC trial: Dutch results. Radiat Oncol. 2020 Feb 18;15(1):41. doi: 10.1186/s13014-020-01487-6. PMID 32070386
- [Derived] Rombouts AJM, Al-Najami I, Abbott NL, Appelt A, Baatrup G, Bach S, Bhangu A, Garm Spindler KL, Gray R, Handley K, Kaur M, Kerkhof E, Kronborg CJ, Magill L, Marijnen CAM, Nagtegaal ID, Nyvang L, Peters FP, Pfeiffer P, Punt C, Quirke P, Sebag-Montefiore D, Teo M, West N, de Wilt JHW; for STAR-TREC Collaborative Group. Can we Save the rectum by watchful waiting or TransAnal microsurgery following (chemo) Radiotherapy versus Total mesorectal excision for early REctal Cancer (STAR-TREC study)?: protocol for a multicentre, randomised feasibility study. BMJ Open. 2017 Dec 28;7(12):e019474. doi: 10.1136/bmjopen-2017-019474. PMID 29288190